CLINICAL TRIAL: NCT00071123
Title: The Functional Neuroanatomy of Emotion Regulation in Major Depressive Disorder (MDD)
Brief Title: Evaluating Brain Responses to Facial Expressions in Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040002; 04-M-0002
Record Dates: First submitted 2003-10-10; First posted 2003-10-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-15

CONDITIONS: Current Major Depressive Disorder; Healthy; Remitted Major Depressive Disorder
Keywords: fMRI; Habituation; Extinction; Amygdala; Emotion; Major Depressive Disorder; Medial Prefrontal Cortex; Backward Masking; Depression; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder, Major; Depression

SUMMARY:
This study will evaluate emotional processing biases in the brain while viewing facial expressions in adults with current or remitted major depressive disorder and healthy volunteers.

DETAILED DESCRIPTION:
The goal of this research is to elucidate the neurophysiological abnormalities associated with processing emotionally valenced stimuli in MDD. Neuroimaging technology has led to the identification of specific abnormalities in the amygdala, ventral striatum and medial prefrontal cortex in response to affective pictures. Much of the knowledge involving these structures in emotion processing has been elucidated through animal models including classical fear conditioning and reversal-learning paradigms. Functional magnetic resonance imaging (fMRI) studies have applied similar techniques in humans to study emotional processing. The amygdala has been shown to play a role in the learning of fear (aversive) conditioning to emotional stimuli, the ventral striatum has been shown to play a role in appetitive conditioning, and areas of the prefrontal cortex are recruited for extinction of conditioned responses. These areas have also been implicated as key structures in the abnormal expression of emotion in MDD. Dysregulation of connections between the amygdala and prefrontal cortex has been hypothesized to influence depressed subjects' tendency to ruminate on emotional events and memories, which may be associated with an inability to properly regulate emotional processing through habituation and extinction mechanisms. Research suggests that depressed individuals have an impaired ability to disengage from or habituate to emotional stimuli perceived as sad.

In addition to studying emotional processing at a conscious, cortical level, significant evidence suggests that many aspects of emotional processing occur below conscious awareness, at a preconscious level. The technique of backward masking assesses the automaticity of emotional processing and responses to affective stimuli. In MDD, backward masking serves to avoid confounding interpretation by the presence of other cognitive processing, which may result from depressed subjects perseverating on emotional stimuli. The proposed study builds on previous fMRI research to investigate neurophysiological differences in the processing of aversively conditioned emotional stimuli in depressed compared to healthy individuals. Using fMRI technology and a variation of the paradigm developed by Morris et al., subjects with MDD will be classically conditioned to the presence of an unmasked specific target face (angry or sad) and the subsequent neural responses to the stimuli will be assessed utilizing the backward masking technique. The BOLD hemodynamic response and rates of habituation and extinction to the faces will be compared between depressed subjects with MDD and healthy controls, currently depressed versus currently remitted subjects with MDD, and MDD subjects pre- and post-antidepressant therapy.

The present amendment proposes to include an additional paradigm in the testing battery. This new paradigm has been extensively examined under different pharmacological manipulations, and in healthy individuals undergoing fMRI but has yet to be examined in patient populations. The task complements the paradigms presently included by extending the research to encompass appetitive as well as aversive emotional processing.

This research will be used to evaluate neural processes involved in emotional dysregulation in MDD and may direct future research to potential therapeutic approaches for the treatment of mood and anxiety disorders with abnormalities in emotional processing.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers (n=65)

Healthy Control Sample (n = 30, phase 1; n = 15, phase 3; n=20, phase 5): Right-handed subjects (ages 18-55) will be selected who have not met criteria for any major psychiatric disorder, have no known first-degree relatives with mood disorders, and have a current score on the Hamilton Depression Rating Scale (HDRS; 17 item) in the not depressed range (less than or equal to 7). Control subjects will be matched to depressed subjects for age, gender, and education.

MDD Samples (n =80)

MDD Sample-Currently Depressed (n = 30, phase 1; n = 15, phase 3; n=20, phase 5): Right-handed subjects (ages 18-55) will be selected with primary MDD currently depressed by DSM-IV criteria for recurrent MDD and current HDRS score in the moderately-to-severely depressed range (greater than or equal to 18).

MDD Sample-Remitted Depressed (n = 15, phase 2): Right-handed subjects (ages 18-50) will be selected with a past history of MDD by DSM-IV criteria.

Healthy Relatives of MDD Subjects (n=45)

Right-handed subjects (ages 18-55) will be selected who have a first-degree relative with MDD but do not themselves meet criteria for a psychiatric disorder. Subjects will be matched to depressed and control subjects for age, gender, and education.

EXCLUSION CRITERIA:

Subjects will be recruited who are drug-na ve or who have not received psychotropic drugs for at least 3 weeks (8 weeks for fluoxetine) prior to scanning. Effective medications will not be discontinued for the purposes of the study. Subjects will also be excluded if they have a) serious suicidal ideation or behavior, b) psychosis to the extent that the ability to provide informed consent is in doubt, c) medical conditions or concomitant medications (see Appendix III) that are likely to influence cerebral blood flow or neurological function including cardiovascular, respiratory, endocrine and neurological diseases, d) a history of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM-IV criteria), e) current pregnancy (as documented by pregnancy testing prior to scanning), f) general MRI exclusion criteria, g) history of non-response to Zoloft or of intolerable or adverse side effects during Zoloft treatment. Additional exclusion criteria applied to control subjects are: a) subjects with a current or past history of other axis I psychiatric conditions, b) subjects with first-degree family members with current or past history of mood disorder.

Subjects beyond age 55 are excluded to reduce the biological heterogeneity encompassed by the MDD criteria, and to reduce the variability of the BOLD signal. Subjects whose first major depressive episodes arose temporally after other major medical or psychiatric conditions will also be excluded, since their functional imaging results generally differ from those reported in primary MDD.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2003-10-09; Study Completion 2010-11-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Morris JS, Buchel C, Dolan RJ. Parallel neural responses in amygdala subregions and sensory cortex during implicit fear conditioning. Neuroimage. 2001 Jun;13(6 Pt 1):1044-52. doi: 10.1006/nimg.2000.0721. PMID 11352610
- [Background] Cahill L, Haier RJ, White NS, Fallon J, Kilpatrick L, Lawrence C, Potkin SG, Alkire MT. Sex-related difference in amygdala activity during emotionally influenced memory storage. Neurobiol Learn Mem. 2001 Jan;75(1):1-9. doi: 10.1006/nlme.2000.3999. PMID 11124043
- [Background] Drevets WC. Prefrontal cortical-amygdalar metabolism in major depression. Ann N Y Acad Sci. 1999 Jun 29;877:614-37. doi: 10.1111/j.1749-6632.1999.tb09292.x. PMID 10415674